CLINICAL TRIAL: NCT02484313
Title: The Effect of Dairy and Non-Dairy Products on Blood Glucose Regulation in Children
Brief Title: The Effect of Snacks on Glycaemic Regulation in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Saint Vincent University (Other)
Collaborators: University of Toronto (Other); IWK Health Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2011-001(2)
Record Dates: First submitted 2015-04-17; First posted 2015-06-29 (Estimated); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Blood Glucose; Energy Intake

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Greek yogurt (Experimental): 25 g available carbohydrates
  Interventions: Other: dietary treatments
- Cookies (Experimental): 25 g available carbohydrates
  Interventions: Other: dietary treatments

INTERVENTIONS:
Other: dietary treatments — commercially available food products

SUMMARY:
Dairy products have a potential to be healthy snack foods for children. The purpose of this project is to investigate the short-term effects of Greek yogurt, a new popular dairy product on the regulation of glucose homeostasis, satiety and energy intake in normal weight and overweight/obese children.

ELIGIBILITY:
Inclusion Criteria:

* The children must be born at full-term within the normal weight range

Exclusion Criteria:

* food sensitivities or allergies, dietary restrictions, health, learning, emotional or behavioural problems, of if children are receiving medication

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2011-11; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
blood glucose | 120 min
  concentration of blood glucose
insulin | 120 min
  concentration of circulating insulin
C-peptide | 120 min
  concentration of circulating C-peptide

SECONDARY OUTCOMES:
Food intake (grams and kcal) | 120 min
  ad libitum food intake at 120 min measured with a test meal (grams consumed converted to kilocalories).
Subjective appetite | 0-120 min
  Four patterns of subjective appetite were measured using 100 mm visual analogue scale (VAS): desire to eat, hunger, fullness, and prospective food consumption at 0 min (immediately before the snack), 15, 30, 45, 60, 90, and immediately before the test meal at 120 min. The average appetite was calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Harvey Anderson, PhD, Principal Investigator — University of Toronto
Locations (1):
- Mount Saint Vincent University, Halifax, Nova Scotia, Canada